CLINICAL TRIAL: NCT06599281
Title: The Importance of Physiotherapy After Separation Surgery in Pygopagus Conjoined Twins
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Ali Demir, Pediatric Physiotherapist, Acıbadem Atunizade Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADemir
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pygopagus Conjoined Twins; Separation Surgery; Pediatric Physiotherapy
Keywords: conjoined twins; pygopagus; physiotherapy; gross motor development; neurodevelopment
MeSH Terms: conditions — Twins, Conjoined | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pygopagus conjoined twins receiving physiotherapy after separation surgery (Other): Physiotherapy was applied to all cases after surgery. The physiotherapy program included neurodevelopmental exercises, balance and proprioception exercises, and stretching exercises.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — The physical therapy program was applied for 3 months, 6 days a week, 2 sessions per day, and an average session duration of 45 minutes. Each neurodevelopmental exercise and proprioceptive exercise was applied for 10 minutes, and stretching exercises were applied for 45 seconds and 3 repetitions. The exercises included functional rotation, sitting with or without arm support, crawling, kneeling, half kneeling, standing up by holding on, and sequencing exercises. Stretching exercises were mostly positional stretches aimed at lateral flexion of the spine.

SUMMARY:
Motor function delays are observed in pygopagus conjoined twins due to limited movement experience and deficits in proprioceptive sense. This study aimed to evaluate the neuromotor development of conjoined twins who acquired independent bodies, lives, and movements as a result of separation surgery, and to examine the effect of postoperative physiotherapy intervention on gross motor function.

DETAILED DESCRIPTION:
The study included two cases of pygopagus conjoined twins who applied for separation surgery at Acıbadem Altunizade Hospital between 2021 and 2022. The twins were 9 months and 21 days old (A1-A2) and 23 months and 11 days old (B1-B2). After separation surgery, a conventional physiotherapy program was administered regularly for 3 months, 6 days a week, with two sessions per day, each lasting 45 minutes. The Bayley-III Developmental Screening Test (DST) was used to evaluate neuromotor development, while the Alberta Infant Motor Scale (AIMS) and the Gross Motor Function Measure-88 (GMFM-88) were used to assess gross motor development. Evaluations were performed preoperatively and at the 3rd postoperative month.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of pygopagus conjoined twins
* Having normal vital signs after separation surgery

Exclusion Criteria:

* Having a diagnosis other than pygopagus conjoined twin
* Abnormal vital signs after separation surgery

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bayley-III Screening Test | 3 months
  The Bayley-III is an individually administered scale that assesses the developmental functions of children aged 1-42 months. It evaluates five domains: cognitive, language, motor, social-emotional, and adaptive behavior. The cognitive (91 items), language (97 items), and motor (138 items) domains are assessed using tasks performed with the child, while the social-emotional and adaptive behavior domains are evaluated based on responses to a questionnaire completed by the caregiver.
  In the cognitive, language, and motor domains, scoring is done as "completed (1)" or "not completed (0)." The Bayley-III provides various scores for each domain, such as raw scores, scale scores, and composite scores. The scale score, derived from standardizing raw scores by age, is a quick and commonly used method in research.
Gross Motor Function Measure-88 (GMFM-88) | 3 months
  The GMFM-88 consists of 88 items and evaluates the child's performance in five different motor skill areas: A. Lying and Rolling (17 items), B. Sitting (20 items), C. Crawling and Kneeling (14 items), D. Standing (13 items) and E. Walking, Running, and Jumping (24 items). Each item in the GMFM-88 is administered by observing the child's natural movements or by giving instructions.
  The items measure the child's ability to perform specific movements. Each movement is scored based on the child's performance, with scores ranging from 0 to 3. 0: Cannot perform the movement, 1: Can partially perform the movement, 2: Can perform the movement independently, 3: Can perform the movement fully and correctly. The scores are summed for each area to obtain a total gross motor function score.
Alberta Infant Motor Scale (AIMS) | 3 months
  The Alberta Infant Motor Scale (AIMS) is an observational assessment used to identify children with delays in motor performance and to provide clinicians and families with information about the child's motor activities. The evaluation of the infant's independent walking and gross motor movements (weight shifting, posture, movements against gravity) takes approximately 20-30 minutes. Movements to be observed are assessed using age-appropriate toys for the infant. During the assessment, the infant continues with spontaneous movements, and postural control is observed while the infant engages in spontaneous motor behaviors.
  The AIMS assessment form contains illustrations of the postures and movements that need to be observed in the infant. It includes 58 items: 21 items in the prone position, 9 items in the supine position, 12 items in the sitting position, and 16 items in the standing position. Each item that the infant can perform is scored as "1," and items that cannot be performed

CONTACTS AND LOCATIONS:
Overall Officials: Gökçen EROL, Principal Investigator — Acıbadem Atunizade Hospital
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.